CLINICAL TRIAL: NCT01867060
Title: Using a Personal Heart Rhythm Monitor (PHRM) to Diagnose Paroxsymal Atrial Fibrillation (PAF) in the Community; and the PREDICT-PAF Substudy - an Investigation of Biomarkers to Detect PAF.
Brief Title: Using a Personal Heart Rhythm Monitor to Diagnose Paroxsymal Atrial Fibrillation in the Community
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HASTE-2
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Paroxysmal Atrial Fibrillation; Stroke
Keywords: Cardiac monitoring; Biomarkers; Transthoracic echocardiography
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Personal Heart Rhythm Monitor (Other): Automated Cardiac Event Recorder in parallel with Personal Heart Rhythm Monitor.
  Interventions: Device: Automated Cardiac Event Recorder; Device: Personal Heart Rhythm Monitor

INTERVENTIONS:
Device: Automated Cardiac Event Recorder — Automated Cardiac Event Recorder to be worn continuously for one week.
  Other Names: 'R. Test Evolution 4' (Novacor).
Device: Personal Heart Rhythm Monitor — Personal Heart Rhythm Monitor to be used twice-daily for three months.
  Other Names: 'Portable ECG monitor HCG-801' (OMRON Healthcare).

SUMMARY:
This propsective study aims to compare the diagnostic yield of a Personal Heart Rhythm Monitor (PHRM) with an automated cardiac event recorder (ACER) to detect paroxysmal Atrial Fibrillation PAF). The investigators hypothesise that the PHRM, used intermittently for 3 months, will detect significantly more cases of PAF than the ACER, used continuously for one week.

A case-control sub-study will identify individuals with confirmed PAF, and matched individuals with no evidence of PAF, to identify potential serum biomarkers for PAF.

A further case-control study will assess markers of left atrial function in patients with PAF and their matched controls.

Another case-control sub-study will determine the significance of frequent Atrial Premature Beats (APBs) in the development of AF over a one year period.

DETAILED DESCRIPTION:
Patients with suspected AF will be initially referred to a community-based, nurse-led Arrhythmia clinic by their General Practitioners over a 15-month period.

All patients will be issued with a one week ACER (the 'R. Test 4 Evolution'), seen as the 'best-practice' investigation for this population group. Participants will also be issued with a PHRM for three months. They will be instructed to take regular twice-daily, 30 second recordings with additional recordings in the event of relevant symptoms. They will return the ACER after one week and the PHRM after 3 months.

A subgroup of participants (target recruitment number = 100) will undergo transthoracic echocardiography. A 40ml venous blood sample will also be taken. Another small subgroup (target recruitment = 20) will be asked to continue twice-daily recordings using the PHRM for a further nine months and will be issued with a repeat one week ACER at study completion.

ELIGIBILITY:
Inclusion Criteria:

* Suspected paroxysmal AF (either palpitations consistent with AF or an irregular pulse)
* 12-lead resting ECG confirming sinus rhythm
* Capacity to consent to study
* English-speaking
* Life expectancy at least one year

Exclusion Criteria:

* Previous diagnosis of AF
* Recent history of syncope
* Recent history of cardiac-sounding chest pain
* A resting ECG suggestive of alternative arrhythmia
* Inability to use the telephone
* Thyrotoxicosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 194 (Actual)
Dates: Start 2013-05; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The diagnostic yield of a Personal Heart Rhythm Monitor (PHRM), used for 3 months, compared to an automated cardiac event recorder (ACER), used for 1 week, to detect all episodes of paroxysmal atrial fibrillation. | 18 months

SECONDARY OUTCOMES:
The diagnostic yield of a Personal Heart Rhythm Monitor (PHRM), used for 3 months, compared to an automated cardiac event recorder (ACER), used for 1 week, to detect prolonged episodes of paroxysmal atrial fibrillation (defined as greater than 12 hours). | 18 months
The sensitivity and specificity of serum biomarkers to detect cases of PAF. | 18 months
The sensitivity and specificity of markers of left atrial function to predict PAF. | 18 months
The development of AF in a cohort confirmed to have frequent atrial ectopic beats (APBs) over a one year period. | 18 months
Adverse events (including stroke/TIA, myocardial infarction, significant bleeding events and death) at six and twelve month intervals. | 30 months
Stroke reduction in the local area | 30 months
  A reduction in stroke burden in the local area will be calculated from estimated stroke risk in individuals identified with AF and from a local registry.
Referrals to secondary care for suspected AF/palpitations | 18 months
  The number of referrals to secondary care for suspected PAF will be analysed.
Participant satisfaction with the devices used in the study. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Howlett, MBChB BSc, Principal Investigator — The Royal Surrey County Hospital; Edward Leatham, MBChB MD, Study Director — The Royal Surrey County Hospital; Chris Fry, BSc PhD, Study Director — The University of Surrey
Locations (1):
- Royal Surrey County Hospital NHS Foundation Trust, Guildford, Surrey, United Kingdom

REFERENCES:
- See also: HASTE charity website — http://www.haste.uk.com